CLINICAL TRIAL: NCT00382603
Title: Clinical Evaluation of the Safety and Efficacy of an Investigational Multi-Purpose Disinfecting Solution Compared to a Marketed Multi-Purpose Solution for Care of Soft Contact Lenses in Symptomatic Patients
Brief Title: Evaluation of an Investigational Multi-Purpose Disinfecting Solution for the Care of Soft Contact Lenses in Symptomatic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-04-09
Record Dates: First submitted 2006-09-28; First posted 2006-09-29 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2006-09

CONDITIONS: Contact Lens Care
Keywords: Contact Lens Care

INTERVENTIONS:
Device: OptiFree Multi-Purpose Disinfecting Solution

SUMMARY:
The objective of the study was to clinically evaluate the safety and effectiveness of a new multi-purpose disinfecting solution for soft contact lenses in patients who experience discomfort with their contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic for contact lens related discomfort at the end of the lens wearing day.
* Successful daily wear of FDA Group IV lenses on a two-week or longer replacement schedule for at least two weeks.
* Use of a multi-purpose solution only as the pre-study care regimen for at least one month (rewetting drops use is also acceptable).
* Successful lens wear for at least 4 hours per day.
* Vision correctable to 20/30.
* Normal eyes - no current ocular abnormalities that prevent successful contact lens wear.
* No corneal surgery within the past 12 months.
* No systemic disease that affects that eye or that could be worsened by the use of contact lenses or solutions.
* No over-the-counter or prescription ocular medication.
* No enrollment in another clinical study within 30 days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 362
Dates: Start 2004-08; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Efficacy:
Ocular Comfort and Symptom Scales
Subject Questions/Subject Likert Questionnaire
Safety:
Slit-lamp Findings - Cornea: Edema, Neovascularization, Infiltrates; Injection, Tarsal Abnormalities and Other Complications
Adverse Events

SECONDARY OUTCOMES:
Corneal Fluorescein Staining (Type and Area)
Lens Surface Evaluation (Lens Deposit and Lens Wettability)
Lens Replacement Incidence and Causality
Corrected Visual Acuity with Study Lenses (Snellen)
Rewetting Drop Frequency
Lens Removal Frequency
Average Lens Wearing Time
Average Uncomfortable Lens Wearing Time

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Napier, Study Director — Alcon Research
Locations (1):
- Highlands Ranch, Highlands Ranch, Colorado, United States